CLINICAL TRIAL: NCT02837367
Title: Use of Nutrigenomic Models for the Personalized Treatment With Medical Foods in Obese People
Acronym: NutriGen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Collaborators: Romania:The National Authority for Scientific Research (Unknown)
Responsible Party: Principal Investigator, Maria Puiu, Professor Dr Maria Puiu, University of Medicine and Pharmacy "Victor Babes" Timisoara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UniversityMedPharmaVBT
Record Dates: First submitted 2016-07-11; First posted 2016-07-19 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Dyslipidemia
Keywords: nutrigenetics; medical foods; obesity; children; adults
MeSH Terms: conditions — Obesity; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Adult intervention (Experimental): The intervention will consist Administration of supplements containing methyl-donors (as capsules) containing: 2 g betaine, 800 ug (micrograms) 5-MTHF (L-5-methyltetrahydrofolate) + 1000 ug (micrograms) Vitamin B12, 500 mg choline bitartrate, 1 g ALA (alfa-linolenic acid), 700 mg EPA (eicosapentaenoic acid), 280 mg DHA (docosahexaenoic acid).
  Every week the participants will receive a weekly amount of supplements, in opaque pharmaceutical-grade plastic bottles, adequately coded. Participants will be instructed to consume the daily amounts in 2-3 administrations, immediately after a meal,for a duration of 3 months
  Interventions: Dietary Supplement: Administration of supplements containing methyl-donors
- Adult placebo (Placebo Comparator): The intervention will consist of the Administration of supplements containing methyl-donors (as capsules) containing inactive ingredients with low glycemic index (usually starch-based), and one capsule containing corn oil (1 g).
  Every week the participants will receive a weekly amount of supplements, in opaque pharmaceutical-grade plastic bottles, adequately coded. Participants will be instructed to consume the daily amounts in 2-3 administrations, immediately after a meal,for a duration of 3 months
  Interventions: Dietary Supplement: Administration of supplements containing methyl-donors
- Children intervention (Experimental): The intervention will consist of the Administration of supplements containing methyl-donors (as syrup) containing: 1 g betaine, 400 ug (micrograms) 5-MTHF (L-5-methyltetrahydrofolate) + 500 ug (micrograms) Vitamin B12, 250 mg choline bitartrate, 0.5 g ALA (alfa-linolenic acid), 700 mg EPA (eicosapentaenoic acid), 140 mg DHA (docosahexaenoic acid).
  Every week the participants will receive a weekly amount of supplements, in opaque pharmaceutical-grade plastic bottles, adequately coded. Participants will be instructed to consume the daily amounts in 2-3 administrations, immediately after a meal,for a duration of 3 months
  Interventions: Dietary Supplement: Administration of supplements containing methyl-donors
- Children Placebo (Placebo Comparator): The intervention will consist of Administration of supplements containing methyl-donors (as syrup) containing inactive ingredients with low glycemic index (usually starch-based), and one capsule containing corn oil (1 g).
  Every week the participants will receive a weekly amount of supplements, in opaque pharmaceutical-grade plastic bottles, adequately coded. Participants will be instructed to consume the daily amounts in 2-3 administrations, immediately after a meal,for a duration of 3 months
  Interventions: Dietary Supplement: Administration of supplements containing methyl-donors
- Adults genetic assessment (No Intervention): Establishing a genetic signature model in the 1-carbon and omega-6/3 fatty acids metabolic pathways, with high predictive value for dyslipidemia and insulin resistance classification in adult people with obesity.
- Children genetic assessment (No Intervention): Establishing a genetic signature model in the 1-carbon and omega-6/3 fatty acids metabolic pathways, with high predictive value for dyslipidemia and insulin resistance classification in children with obesity.

INTERVENTIONS:
Dietary Supplement: Administration of supplements containing methyl-donors — Administration of supplements containing methyl-donors: betaine, 5-MTHF (L-5-methyltetrahydrofolate), Vitamin B12, choline bitartrate, ALA (alfa-linolenic acid), EPA (eicosapentaenoic acid), DHA(docosahexaenoic acid)
  Arms: Adult intervention; Adult placebo; Children Placebo; Children intervention

SUMMARY:
The NutriGen project will be using nutrigenomic methods to determine the effectiveness of treatments with specific dietary foods, on the basis of genetic risk predisposition (genetic signature) of obese individuals.

DETAILED DESCRIPTION:
NutriGen project specific aim 1. Establishing a genetic signature model, involved in the donation of methyl groups and unsaturated omega-6/3 fatty acids metabolism, with a high predictive value for classification of dyslipidemia and insulin resistance in obese subjects.

1. Establishing a genetic signature model in obese adults with dyslipidemia.
2. Establishing a genetic signature model in obese children with insulin resistance. c. Establishing a correlation between blood/plasma concentrations of the relevant metabolites, genetic signatures and dyslipidemia profile of adults, and respectively a profile for insulin resistance in obese children.

NutriGen project specific aim 2. Determining the efficacy of a dietary food specific treatment, which is also correlated with a genetic signature (nutrigenomics), based on the correlations defined in objective 1:

1. Implementation of a treatment with dietary foods (for adults), in the presence/absence of other already prescribed treatments;
2. Implementation of a treatment with dietary foods (for children), in the presence/absence of other already prescribed treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adults: between 18 and 70 years old; obesity present as defined by body mass index (BMI) ≥30 kg/m2 and by abdominal circumference ≥84 cm (women), and ≥90 cm (men); dyslipidemia present as defined by: serum Cholesterol ≥200 mg/dl, HDLc ≤50 mg/dl (women) or ≤40 mg/dl (men), serum Triglycerides ≥150 mg/dl, or present treatment for dyslipidemia (e.g. statins, fibrates, omega-3 fatty acids, cholestyramine, ezetimibe).
* Children: age between 7 and 18 years old; BMI >+2SD WHO reference

Exclusion Criteria:

* Adults: diagnosed for any type of cancer, or medical history of cancer; any auto-immune disease; any psychiatric disorder; blood coagulation disorders; history of drug abuse; alcohol abuse evaluated using AUDIT-C.
* Children: the above exclusion criteria for adults; familial hypercholesterolemia; endocrine-induced obesity (Cushing syndrome, hypothyroidism, growth hormone deficit), hypothalamus-induced obesity (Babinski-Fröhlich syndrome), genetic syndromes (Prader-Willi, achondroplasia, Bardet-Biedl, Fanconi, Turner, etc.); deposition diseases (glycogenosis, lipomatosis); personal history for: convulsive disorders, nephrotic syndrome, or asthma that necessitated corticoid treatment.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Lipid profile | 3 years
  HDL-cholesterol (HDLc), LDL-cholesterol (LDLc), triglycerides (TG)

SECONDARY OUTCOMES:
Insulin sensitivity | 3 years
  HOMA-IR

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Niculescu, MD, PhD, Principal Investigator — University of Medicine and Pharmacy "Victor Babes" Timisoara
Locations (2):
- Romania (2):
  - Clinica II Pediatrie Bega, Timișoara, Timiș County
  - Spitalul Judetean Timisoara; Centrul de Diabet, Timișoara, Timiș County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corbin KD, Abdelmalek MF, Spencer MD, da Costa KA, Galanko JA, Sha W, Suzuki A, Guy CD, Cardona DM, Torquati A, Diehl AM, Zeisel SH. Genetic signatures in choline and 1-carbon metabolism are associated with the severity of hepatic steatosis. FASEB J. 2013 Apr;27(4):1674-89. doi: 10.1096/fj.12-219097. Epub 2013 Jan 4. PMID 23292069
- [Derived] Chirita-Emandi A, Serban CL, Paul C, Andreescu N, Velea I, Mihailescu A, Serafim V, Tiugan DA, Tutac P, Zimbru C, Puiu M, Niculescu MD. CHDH-PNPLA3 Gene-Gene Interactions Predict Insulin Resistance in Children with Obesity. Diabetes Metab Syndr Obes. 2020 Nov 19;13:4483-4494. doi: 10.2147/DMSO.S277268. eCollection 2020. PMID 33239899
- [Derived] Serban CL, Sima A, Hogea CM, Chirita-Emandi A, Perva IT, Vlad A, Albai A, Nicolae G, Putnoky S, Timar R, Niculescu MD, Puiu M. Assessment of Nutritional Intakes in Individuals with Obesity under Medical Supervision. A Cross-Sectional Study. Int J Environ Res Public Health. 2019 Aug 22;16(17):3036. doi: 10.3390/ijerph16173036. PMID 31443343